CLINICAL TRIAL: NCT03653754
Title: Growth and Body Composition in Children With Disabilities and Typically Developing Children
Brief Title: Growth and Body Composition in Children
Status: Completed | Type: Observational
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Bo Young Hong, Associate professor, The Catholic University of Korea
Other Study IDs: VC17ONSI0200
Record Dates: First submitted 2018-07-24; First posted 2018-08-31 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Growth; Child Development; Disability, Developmental
Keywords: growth; Body Composition
MeSH Terms: conditions — Developmental Disabilities | interventions — Body Composition

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- typically developing: Intervention: Measurement of growth and body composition. Growth (height, body weight), and body composition was measured at school.
  Interventions: Diagnostic Test: Measurement of growth and body composition
- neurodisabilities: Intervention: Measurement of growth and body composition. Growth (height, body weight), and body composition was measured at school.
  Interventions: Diagnostic Test: Measurement of growth and body composition

INTERVENTIONS:
Diagnostic Test: Measurement of growth and body composition — Growth (height and body weight), and body composition were measured. For the body composition, Inbody 770 and Inbody S10 were used.
  Other Names: Using Inbody 770, Inbody S10

SUMMARY:
This study is planned to measure and compare body composition indexes and growth between typically developing children and those with disabilities in South Korea for understanding the nutritional and growth status.

DETAILED DESCRIPTION:
* Inclusion criteria for typically developing children

  1. typically developing children in 5th and 6th grades of elementary schools
  2. children whose parents checked the agreement form distributed by schools
* Inclusion criteria for children with disabilities

  1. children and adolescent who are in special schools
  2. children whose parents checked the agreement form distributed by schools
  3. children who were able to cooperate during the body composition analysis
* Exclusion criteria for both groups

  1. those whom do not have written informed consent
  2. who are not able to stay calmly during the body composition analysis
* All measurements done at two elementary schools on the day of the annual physical examination
* Measurement of height and body weight for growth
* Measurement of body composition index: Inbody 770 and Inbody S10, body composition analyzers

ELIGIBILITY:
Inclusion Criteria:

* Those who agreed to participate both parents and a child
* Typically developing children: among the 5th and 6th grade of two elementary schools.
* Children with neurodevelopmental disabilities: among the students in a special school.

Exclusion Criteria:

* Who do not want to participate
* Who are not possible to do the Inbody examination

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 1. Typically developing children who are in the 5th and 6th grades of elementary schools
  2. Children with neurodevelopmental disabilities in a special school
Sampling Method: Non-Probability Sample
Enrollment: 428 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-11-29 (Actual)

PRIMARY OUTCOMES:
BW | through study completion, an average of 1.5 month
  body weight (kg)

SECONDARY OUTCOMES:
skeletal muscle mass (kg) | through study completion, an average of 1.5 month
  skeletal muscle mass measured by body composition analyzers (Inbody 770 and Inbody S10)
fat mass (kg) | through study completion, an average of 1.5 month
  fat mass measured by body composition analyzers (Inbody 770 and Inbody S10)
height | through study completion, an average of 1.5 month
  height

CONTACTS AND LOCATIONS:
Overall Officials: Bo Young Hong, MD, PhD, Principal Investigator — St. Vincent's hospital, The Catholic University of Korea
Locations (1):
- St. Vincent's Hospital, The Catholic University of Korea, Suwon, South Korea

IPD SHARING:
Plan to Share IPD: No